CLINICAL TRIAL: NCT00642772
Title: Pilot Study of Group Physical Therapy for Knee Osteoarthritis
Brief Title: Group Physical Therapy for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SHP 08-180
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Veterans; Physical Therapy; Health Services Research
MeSH Terms: conditions — Osteoarthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Physical Therapy (Experimental): 12-week group-based program of physical therapy. Participants will meet approximately every other week for a total of 6 visits. The group sessions will include education about appropriate self-care for knee osteoarthritis and instructions and participation in group exercises. Participants will also be instructed in a home exercise program.
  Interventions: Other: Group Physical Therapy

INTERVENTIONS:
Other: Group Physical Therapy — 12-week group-based program of physical therapy. Participants will meet approximately every other week for a total of 6 visits. The group sessions will include education about appropriate self-care for knee osteoarthritis and instructions and participation in group exercises. Participants will also be instructed in a home exercise program.

SUMMARY:
Osteoarthritis (OA) is a common cause of pain and disability. Physical therapy is a key part of treatment for OA, but VA Medical Centers are often limited in their capacity to provide physical therapy services for veterans with knee OA. The goal of this study is to perform a preliminary work on a group-based physical therapy program for veterans with knee osteoarthritis (OA), in preparation for a larger project. This work will allow us to assess the feasibility of conducting group-based physical therapy program and to plan a larger grant submission based on the findings of this initial study. We hypothesize that the group-based program will be feasible to administer and will result in improved pain and function.

DETAILED DESCRIPTION:
Background / Rationale: Osteoarthritis (OA) is the one of the most common chronic conditions among veterans, and over half of VA health care users with OA report being limited in their daily activities because of joint symptoms. Physical therapy and ongoing exercise help to reduce pain and improve physical function. However, the majority of veterans with OA are physically inactive. Furthermore, physical therapy appointments in the VA health care system are a limited resource, with demand often exceeding supply, resulting in long wait periods and a limited number of visits (1 or 2) per patient. Extending physical therapy services to a larger number of veterans with OA, in a cost effective manner, may play a key role in improving outcomes in this large patient group. Objective: The objective of this pilot study is to perform preliminary evaluation of group-based physical therapy program for veterans with knee OA, in preparation for a larger grant submission. This pilot work will allow us to assess the feasibility of group-based sessions, refine the intervention session components as needed, assess the planned recruitment and enrollment methods, estimate the number of potentially eligible veterans at the Durham VAMC, and conduct sample size and power analyses for a larger clinical trial. Methods: All participants will be involved in a 12-week group-based physical therapy program, with study measures being obtained at baseline and immediately following program completion. Participants will be Durham VAMC patients with symptomatic knee OA. Our goal is to enroll 20 participants who complete the program and follow-up measures, but we may recruit up to 25 participants total, if some participants drop out of the program before completion. Participants will attend group physical therapy sessions bi-weekly for twelve weeks (total of six visits), with each session lasting approximately one hour. Two study team members, a licensed physical therapist and research assistant with training in exercise for knee OA, will lead each session. The research assistant will lead group exercises, and the physical therapist will assess the progress and monitor for any potential problems or special needs of individual patients. During the first 10-15 minutes of each group session, one study team member will talk with participants about a topic related to OA care, such as joint protection, weight management, joint injections and surgery, and stress management. The remainder of the session will involve group warm-up / stretching exercises, then a series of strengthening exercises tailored for patients with knee OA. Participants will also be instructed to perform stretching exercises daily and strengthening exercises three times total each week. Primary outcome measures will be self-reported pain and function. Statistical analyses will compare pre- and post-intervention pain and function, including effect size calculations to assist with sample size estimates for a larger study. Impact: This study is significant because it examines a novel health services delivery method for improving outcomes among patients with OA - a highly prevalent condition that is also one of the main causes of pain among veterans. Specifically, this pilot study is a key first step toward examining the efficacy and cost-effectiveness of a method for delivering physical therapy services to a larger number of veterans with OA. This delivery method could also be applied to other common orthopedic and neurologic conditions that require physical therapy service.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic Evidence of Knee Osteoarthritis and a Clinician's Diagnosis
* Current knee symptoms

Exclusion Criteria:

* Presence of other rheumatological conditions (such as rheumatoid arthritis and fibromyalgia) - Other health-related problem that would prevent safe participation in a physical therapy program - Currently undergoing physical therapy for knee OA, participation in another interventional study, scheduled or on waiting list for joint replacement surgery, resident of nursing home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Physical Therapy: Group Physical Therapy Intervention
  Group Physical Therapy: 12-week group-based program of physical therapy. Participants will meet approximately every other week for a total of 6 visits. The group sessions will include education about appropriate self-care for knee osteoarthritis and instructions and participation in group exercises. Participants will also be instructed in a home exercise program.
Period: Overall Study
Arm/Group | Group Physical Therapy
Started | 24
Completed | 14
Not Completed | 10
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Group Physical Therapy
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: Self-report measure of pain (5 items), stiffness (2 items) and function (17 items) in lower extremity osteoarthritis. All items were measured on a 5-point likert scales, with higher scores indicating worse pain, stiffness, or functional limitations. Total WOMAC score ranges from 0-96.
Time Frame: Baseline and Following 12-Week Intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Physical Therapy
Number analyzed (Participants) | 14
units on a scale
  Baseline Score | 43.3 (14.6)
  12-Week Score | 34.1 (16.0)

ADVERSE EVENTS:
Time Frame: During 12 week intervention period for each participant
Arm/Group | Group Physical Therapy
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No